CLINICAL TRIAL: NCT01708759
Title: The Value of Admission Serum Il-8 Monitoring and the Detection of IL8 (-251 A/T) Polymorphism in Critically Ill Patients
Brief Title: IL8 Monitoring and Its Correlation With 251-gene Polymorphism
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman Abd Al-maksoud Yousef, Assistant professor of Anesthesiology, Tanta University
Other Study IDs: 1380/09/12
Record Dates: First submitted 2012-10-12; First posted 2012-10-17 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Sepsis; Systemic Inflammatory Response Syndrome
Keywords: Serum Il-8; IL8 polymorphism; critically ill patients
MeSH Terms: conditions — Sepsis; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Sepsis: Forty patients developed septic complication during ICU stay (sepsis group).
- SIRS: Forty patients were critically ill without evidence of infectious organism (SIRS group).

SUMMARY:
One hundred eighty critically ill African adult intensive care patients divided into two groups, eighty septic critically ill patients (sepsis group) while, eighty non-septic critically ill patients (SIRS) group. Admission serum IL-8 was measured in both sepsis and SIRS groups. IL-8 (-251A/T) polymorphism was detected in sepsis and SIRS groups.

DETAILED DESCRIPTION:
A total of one hundred eighty African patients (97men and 83 women) were included in the study. Eighty patients developed septic complication during ICU stay (sepsis group). Eighty patients were critically ill without evidence of infectious organism (SIRS group). Patients received anti-inflammatory drugs or corticosteroids before admission, who had immunosuppressive illness, who had chronic organ failure; who had received massive blood transfusion; those with radiation therapy, previous organ transplantation were excluded from the study. At admission, the patient's age, sex, height and weight were recorded. These data include the following: clinical status; sequential organ failure assessment (SOFA) score; temperature; heart rate; respiratory rate; blood pressure; central venous pressure; laboratory analysis (complete blood count, blood urea nitrogen, blood sugar, serum sodium, potassium, calcium, aspartate aminotransferase, alanine aminotransferase, prothrombin time, albumin and CRP) and arterial blood gas analysis. Routine cultures of blood, urine and suspected sites were obtained to determine the presence of infection. We attempted to maintain the patient hemoglobin level at 10-12g/dl and central venous pressure at 8-12 cmH2o. If needed, blood products, intravascular fluid replacement and inotropic and/or vasopressor agents were administered. Each day the attending physician in the ICU evaluated all the study patients for sepsis, severe sepsis, or septic shock.

ELIGIBILITY:
Inclusion Criteria:

Adults patients with clinical diagnosis of sepsis or systemic inflammatory response syndrome.

Exclusion Criteria:

Patients received anti-inflammatory drugs or corticosteroids before admission, patients who had immunosuppressive illness ie. AIDS, patients with chronic liver failure, patients with renal failure, patients with respiratory failure ; patients received massive blood transfusion; patients with radiation therapy, patients with organ transplantation .

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: A total of eighty African patients (47men and 33 women) were included in the study. Forty patients developed septic complication during ICU stay (sepsis group). Forty patients were critically ill without evidence of infectious organism (SIRS group).
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2012-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Serum Interlukin-8 | At intensive care admission. Patients will be followed for at least 2 weeks
  Serum level of IL-8 was determined by quantitative sandwich enzyme immunoassay (R&D Systems, Inc., Minneapolis, MN, USA) according to the manufacturer's instructions. The intensity of the colour was measured at 490 nm for IL-8.

SECONDARY OUTCOMES:
Interlukine-8polymorphism at 251 A/t | At ICU admission. Patients will be followed for at least 2weeks.
  About 4ml blood is withdrawn in EDTA-tubes and the genomic DNA was extracted. Concentration of the extracted DNA was then measured by UV spectrophotometry at 260& 280 nm and run on agaros gel electrophoresis 2% for detection of purity. Molecular detection of the (-251 A/T) polymorphism in the IL-8gene was achieved by restriction fragment length polymorphism typing.

CONTACTS AND LOCATIONS:
Overall Officials: Ayman A Yousef, MD, Principal Investigator — Assistant professor os Anesthesia and ICU, Faculty of Medicine, Tanta university
Locations (1):
- Faculty of Medicine ,Tanta University., Tanta, Algharbiya, Egypt

REFERENCES:
- [Background] Sutherland A M, Russell J A. Issues with polymorphism analysis is sepsis. Clinical infectious diseases 2005; 41; S369-402. Winning J, Claus RA, Huse K, Bauer M. Molecular biology on the ICU from understanding to treating sepsis. Minerva Anestesiol 2006; 72:255-67. Hull J, Thomson A, Kwiatkowski D:Association of respiratory syncytial virus broncholitis with the interleukin-8 gene region in UK families. Thorax 2000, 55: 1023-1027. Gyulai Z, Klausz G, Tiszai A, Lenart Z, Kasa IT, Lonovics J, Mandi Y. Genetic polymorphism of interleukin-8 (IL-8) is associated with Helicobacter pylori induced duodenal ulcer. Eur Cytokine Netw 2004, 15:353-358.